CLINICAL TRIAL: NCT03014908
Title: Metabolic Profiling of Type 1 Diabetes Mellitus in Children and Adolescents: a Case-control Study
Brief Title: Metabolic Profiling of Type 1 Diabetes Mellitus in Children and Adolescents
Acronym: T1DM
Status: Completed | Type: Observational
Sponsor: Hasselt University (Other)
Collaborators: Jessa Hospital (Other)
Responsible Party: Principal Investigator, Peter Adriaensens, professor (hoogleraar), Hasselt University
Other Study IDs: LCRP-obesitas
Record Dates: First submitted 2016-12-12; First posted 2017-01-09 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2017-01

CONDITIONS: Type1diabetes
Keywords: Type 1 diabetes; 1H-NMR spectroscopy; Metabolomics; Pediatrics
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood plasma for proton-NMR spectroscopy

GROUPS / COHORTS (2):
- NMR-T1DM: type 1 diabetic children and adolescents
  Interventions: Other: Blood sampling
- NMR-C: non-diabetic children and adolescents
  Interventions: Other: Blood sampling

INTERVENTIONS:
Other: Blood sampling — Determine the metabolic phenotype of blood plasma by proton-NMR spectroscopy

SUMMARY:
The aim of this study was to look for discriminating variation in the concentrations of small-molecule metabolites in the plasma of T1DM children compared with non-diabetic matched controls using proton nuclear magnetic resonance (1H-NMR)-based metabolomics.

DETAILED DESCRIPTION:
Type 1 diabetes mellitus (T1DM) is one of the most common pediatric diseases and its incidence is rising in many countries. Recently, it has been shown that metabolites other than glucose play an important role in insulin deficiency and the development of diabetes. The aim of this study was to look for discriminating variation in the concentrations of small-molecule metabolites in the plasma of T1DM children compared with non-diabetic matched controls using proton nuclear magnetic resonance (1H-NMR)-based metabolomics.

This cross-sectional study was set-up to examine the metabolic profile in fasting plasma samples from 7 T1DM children and 7 non-diabetic controls aged 8 to 18 years, and matched for gender, age and BMI. The obtained plasma 1H-NMR spectra were rationally divided into 110 integration regions, representing the metabolic phenotype. These integration regions reflect the relative metabolite concentrations and were used as statistical variables to construct (train) a classification model in discriminating between T1DM patients and controls.

ELIGIBILITY:
Inclusion Criteria:

* aged between 8 and 18
* normal-weight according to the International Obesity Task Force (IOTF) BMI criteria
* fasted for at least 8 hours.

Exclusion Criteria:

* lipid-lowering drugs or other medication

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: from 7 T1DM children and 7 non-diabetic controls aged 8 to 18 years, and matched for gender, age and BMI
Sampling Method: Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2014-01; Primary Completion 2014-09 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Metabolic phenotype of type 1 diabetes mellitus | 10 months
  Significant metabolic changes in blood plasma of type 1 diabetic patients compared with control subjects

CONTACTS AND LOCATIONS:
Overall Officials: Peter Adriaensens, PhD, Principal Investigator — Institute of Material Research, Hasselt University; Guy Massa, PhD, MD, Study Chair — Jessa Ziekenhuis Hasselt; Wanda Guedens, PhD, Study Chair — Hasselt University; Evelyne Louis, PhD, Study Chair — Hasselt University; Jean-Paul Noben, PhD, Study Chair — Hasselt University; Liene Bervoets, PhD, Study Chair — Hasselt University
Locations (1):
- Hasselt University, Hasselt, Limburg, Belgium

REFERENCES:
- [Background] Beckonert O, Keun HC, Ebbels TM, Bundy J, Holmes E, Lindon JC, Nicholson JK. Metabolic profiling, metabolomic and metabonomic procedures for NMR spectroscopy of urine, plasma, serum and tissue extracts. Nat Protoc. 2007;2(11):2692-703. doi: 10.1038/nprot.2007.376. PMID 18007604
- [Background] Brugnara L, Mallol R, Ribalta J, Vinaixa M, Murillo S, Casserras T, Guardiola M, Vallve JC, Kalko SG, Correig X, Novials A. Improving Assessment of Lipoprotein Profile in Type 1 Diabetes by 1H NMR Spectroscopy. PLoS One. 2015 Aug 28;10(8):e0136348. doi: 10.1371/journal.pone.0136348. eCollection 2015. PMID 26317989
- [Background] Lanza IR, Zhang S, Ward LE, Karakelides H, Raftery D, Nair KS. Quantitative metabolomics by H-NMR and LC-MS/MS confirms altered metabolic pathways in diabetes. PLoS One. 2010 May 10;5(5):e10538. doi: 10.1371/journal.pone.0010538. PMID 20479934